CLINICAL TRIAL: NCT03298425
Title: The Use of Neuromuscular Electrical Muscle Stimulation With Pelvic Fracture Rehabilitation: A Double Blind, Placebo Controlled, Randomised Control Trial
Brief Title: The Use of NMES With Pelvic Fracture Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BartsLondonNHS
Record Dates: First submitted 2015-07-08; First posted 2017-10-02 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-06

CONDITIONS: Fractures, Closed
MeSH Terms: conditions — Fractures, Closed

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment NMES (Active Comparator): Patients allocated to the NMES group will be given an information booklet on NMES machines. The Cefar Compex three electrical stimulator will be used. Participants are expected to use the NMES machine for half an hour and complete bed exercises twice daily. Patients should relax during the NMES as completing both does not demonstrate better results, due to unsynchronised activation of the NMES (Gregory & Bickel, 2005). Using the machine once daily will allow for the recovery of the muscle. A voluntary contraction would normally be 20-30Hz but due to the high intensities of the NMES (35-75Hz) it can cause muscle fatigue (Maffiuletti, 2011).
  Interventions: Device: Treatment NMES
- Placebo NMES (Placebo Comparator): The placebo group will act as the control group. They will be expected to complete the same regime as previously described above, however these machines will be on TENS setting (80-100Hz) as even low Hz can trigger motor stimulation (Paillard 2008). This setting is designed as a sensory stimulus therefore will have no effects on muscle strength however the patient will feel a small twitch sensation. This setting is not painful and will have no effect on muscle fatigue. The patient will not be expected to complete the bed exercises and the TENS session together.
  Interventions: Device: Placebo NMES

INTERVENTIONS:
Device: Treatment NMES — Muscle stimulation to reproduce an active muscle contraction. CE marked used for intended purpose.
  Arms: Treatment NMES
Device: Placebo NMES — TENS machine to mimic an active muscle contraction. CE marked used for intended purpose.
  Arms: Placebo NMES

SUMMARY:
The purpose of the study is to investigate if using an electrical stimulation machine to see if it can help strengthen the muscles around the hip during the first three months post pelvic fracture will help with the early stages of rehabilitation. Electrical stimulation is a treatment machine that uses an electrical current to cause a single muscle or a group of muscles to contract. This contraction helps strengthen injured muscles and helps with the healing process. It can also help with pain relief by blocking pain signals from the brain.

After a pelvic fracture they are surgically fixed and will be advised not to put any weight on the operated leg for 10 weeks. During this time hip muscles become very weak as they will not be used as much as normal. Bed exercises can help keep muscle strength but this study would like to try using electrical stimulation machines alongside bed exercises to see if it can improve muscle strength even more. Electrical stimulation machines are already used by rehabilitation. Electrical stimulation is a treatment machine that uses an electrical current to cause a single muscle or a group of muscles to contract. This contraction helps strengthen injured muscles and helps with the healing process. It can also help with pain relief by blocking pain signals from the brain.

After a pelvic fracture they are surgically fixed and will be advised not to put any weight on the operated leg for 10 weeks. During this time hip muscles become very weak as they will not be used as much as normal. Bed exercises can help keep muscle strength but this study would like to try using electrical stimulation machines alongside bed exercises to see if it can improve muscle strength even more. Electrical stimulation machines are already used by patients to increase muscle strength.

Participants will be put into one of two groups, both groups will be given an electrical stimulation machine but one will be on a placebo setting. Participants will need to use the machine twice a day along with their bed exercises and will need to fill in a diary when and how many times the machine has been used for 10 weeks until their 12 week appointment with the orthopaedic consultant. The participants weight bearing status will change and they will be asked to perform a muscle strength test on both the operated and nonoperated leg. They will also have their walking quality assessed. The results will compare both groups for muscle strength and walking changes.

DETAILED DESCRIPTION:
All subjects who wish to enter the study will be fully screened and consented by the Chief Investigator, or an appropriate delegate. The Royal London is the largest major trauma centre in London and fixes more pelvic fractures than any other hospital. The orthopedic team will surgically fix between two and six pelvic fractures per week which should meet the inclusion criteria. Pelvic fractures are surgically fixed and then will be instructed to put no weight through the operated limb for 10-12 weeks by the orthopedic consultant. The physiotherapist will give the patient a bed exercise programme day one post operation as per standard practice which consists of hip range of movement exercises and gentle strengthening exercises for muscles around the hip and thigh.

The chief investigator will be part of the patient's normal healthcare team and will identify eligible participants. The participants will be recruited one week post operation to give the patient time to recover from their surgery but not allow for loss in muscle mass. The research assistant will approach the participant 24 hours prior to this and explain the demands of the study and what it will involve allowing the participant 24 hours to discuss this with family members.

After the 24 hour period the chief investigator will also be present to answer any questions about the study. The participant will be expected to provide written informed consent and will be expected to sign the treatment contract which outlines the responsibilities of the participant and the chief investigator. On discharge a six week follow up appointment in fracture clinic will be arranged in which both the consultant and chief investigator will be present to complete the EQ5D questionnaire and monitor compliance within the first six weeks of the intervention. At 10 weeks the participant will have a further fracture clinic appointment in which they are expected to bring back the machine and make a short journey to the human performance laboratory and Queen Mary's University to complete their gait analysis and strength testing along with a further EQ5D questionnaire, this will be the end of the study and the participants are free to leave.

Randomisation procedure

Simple random sampling will be used with a free randomisation computer programme (www.sealedenvelopes.co.uk). When the patient has consented to the study the chief investigator will enter the participant unique study number into the website whilst the participant can read the patient information sheet and treatment contract and it will randomly allocate into treatment (NMES) or placebo (TENS) group. If a participant withdrew from the study a new participant could not replace this participant but be randomly allocated into a group as a new patient.

Blinding/ Emergency unblinding

The independent assessor will be blinded to participant allocation when testing at 10 weeks for both the gait analysis and peak torque measurements. All participants will be blinded to group allocation and will all be given identical machines on different settings. The principle investigator will complete the randomisation procedure and will be aware of group allocation for monitoring and safety purposes.

Treatment/intervention plan and rationale

Patients allocated to the NMES group will be given an information booklet on NMES machines and the principle researcher will explain and demonstrate how to use the machines. The Cefar Compex three electrical stimulator will be used and demonstrates valid results from previous studies (Billot et al 2010., Gondin et al 2005., and Maffiuletti et al., 2002).

Participants are expected to use the NMES machine for half an hour and complete bed exercises twice daily. They will be activating two of their muscles at the same time and will not be expected to complete the bed exercises and NMES together. Patients should relax during the NMES as completing both does not demonstrate better results, due to unsynchronised activation of the NMES (Gregory & Bickel, 2005). Using the machine once daily will allow for the recovery of the muscle. A voluntary contraction would normally be 20-30Hz but due to the high intensities of the NMES (35-75Hz) it can cause muscle fatigue (Maffiuletti, 2011).

Participants will use the muscle reinforcement rehabilitation protocol below which increases from 4Hz to 85Hz allowing slow and fast twitch muscle fibre recruitment. This protocol is used for participants who have had minimal loss of muscle bulk and starts with small currents and slowly builds up as the patient becomes accustom to the sensation of the machine. Patients are expected to increase the intensity, as higher intensity can increase activation of more muscle fibres (Stevens-Lapsley et al, 2012).

Additional treatment/ interventions

The placebo group will act as the control group. They will be expected to complete the same regime as previously described above, however these machines will be on TENS setting (80-100Hz) as even low Hz can trigger motor stimulation (Paillard 2008). This setting is designed as a sensory stimulus therefore will have no effects on muscle strength however the patient will feel a small twitch sensation. This setting is not painful and will have no effect on muscle fatigue. The patient will not be expected to complete the bed exercises and the TENS session together.

Experts within orthopedic rehabilitation concluded a 20% difference between operated and non-operated post intervention would be of clinical relevance. A randomized feasibility study was completed previously in which the results were used to calculate a power calculation for this specific trial. The value of 0.25 represents the standard deviation achieved when comparing the NMES and the placebo group in the previous study. The 0.2 is 20% calculated into a ratio which is needed to achieve clinical relevance. This power calculation indicates 25 participants are needed for each group to achieve statistical significance 50 participants in total. The orthopedic team will surgically fix between two and six pelvic fractures per week which should meet the inclusion criteria. Dropout rates will be small as it is a six week intervention. Patients will receive weekly phone calls and text reminders monitoring compliance.

N= (1.96+0.84)2 x 2 x 0.252 0.22 = 25 per group (50 in total)

0.2/ 0.25 = the standard deviation achieved when comparing treatment to placebo in peak torque differences

0.2 = is the ratio / 20% difference between the treatment and placebo group in abductors

An independent experimental design using an independent test will be suitable to assess the data for this study. Both the placebo and NMES group will have different interventions and will therefore not be measured using a pre and post design. Due to the adequate sample size it will be appropriate to use a parametric statistical test. A Paired T-test will be used to analyse the data from the EQ5D questionnaire as they are taken at six and 12 weeks during the intervention with the same participants.

A Spearman's rank correlation test will be used to compare changes with compliance levels in both bed exercises and NMES use in the NMES group and compared to the changes in peak torque to assess the relationship between the two variables. The same will be completed between the intensity level of the NMES and the changes in peak torque within the NMES group. Variables can be seen in table format below:

ELIGIBILITY:
Inclusion Criteria:

* Patients who can give written informed consent
* Patients with surgically fixed pelvic fractures who are TTWB for up to 10-12 weeks
* Patients with associated injuries considered for example fractured upper limb however their recovery must be within six weeks when they start the intervention.
* Males and females between 18-70 years old
* Patients able to comply and complete the electrical stimulation machine and complete both bed exercises and NMES twice daily.

Exclusion Criteria:

* Patients with current or previous mental health, chronic pain or previous injury which may affect participation.
* Any complex lower limb injury in either limb unless fixed and cleared six weeks post injury.
* Severe kidney injuries which are ongoing will not considered following a case of rhabdomyolysis induced by excessive NMES (Guarascio et al, 2004).
* Patients who may be pregnant
* Patients who suffer from sensitivity problems for the skin
* Patients who may have an abdominal or Inguinal hernia
* Patients with arterial circulation disorders of the lower limb
* Patients with pacemakers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Muscle strength in peak torque between treatment and placebo group | 10 weeks
  HUMAC isokinetic machine

SECONDARY OUTCOMES:
Gait analysis | 10 weeks
  to assess participants gait analysis post intervention - Using gait analysis equipment at a gait analysis lab
EQ5D questionnarrie | 10 weeks
  pre and post intervention EQ5D scores

CONTACTS AND LOCATIONS:
Overall Officials: Jessica A Rich, MRes, Principal Investigator — Barts Health